CLINICAL TRIAL: NCT04854993
Title: Recovery From Deep Neuromuscular Blockade Using Different Sugammadex Doses in Elderly Patients Undergoing Laparoscopic Robot-assisted Prostatectomy: a Prospective, Randomized, Double-blind Clinical Trial
Brief Title: Recovery From dNMB Using Different Sugammadex Doses in Elderly Patients Undergoing Robot-assisted Prostatectomy
Acronym: RECIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3764; 2020-004704-34 (EudraCT Number)
Record Dates: First submitted 2021-04-14; First posted 2021-04-22 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer; Neuromuscular Blockade
Keywords: sugammadex; elderly; recovery time; robotic surgery
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient as well as the investigator (care provider) who will administer the different blinded sugammadex dosage and collect postoperative data will be blinded to the group allocation. The randomization and preparation of the drug will be performed by the unblinded staff of hospital experimental pharmacy who will carry out the randomization with a 1: 1 ratio and will assign the different dose to each patient. The drug will be prepared in a shielded pre-filled syringe in order to maintain blindness. In case of emergency, the pharmacy staff will immediately open the randomization code of interest disclosing the group assignment (sugammadex dose).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Increased dose of sugammadex (Experimental): A dose of 6 mg/kg of sugammadex will be given intravenously for deep neuromuscular block reversal at the end of surgery
  Interventions: Drug: Sugammadex 6 mg/kg
- Standard dose of sugammadex (Active Comparator): A dose of 6 mg/kg of sugammadex will be given intravenously for deep neuromuscular block reversal at the end of surgery
  Interventions: Drug: Sugammadex 4 mg/kg

INTERVENTIONS:
Drug: Sugammadex 6 mg/kg — i.v. injection of an increased (by 50%) dose of sugammadex to reverse dNMB
  Other Names: MK-8616
  Arms: Increased dose of sugammadex
Drug: Sugammadex 4 mg/kg — i.v. injection of a standard dose of sugammadex to reverse dNMB
  Other Names: MK-8616
  Arms: Standard dose of sugammadex

SUMMARY:
The aim of this prospecive randomized study is to evaluate the effects of a dose of sugammadex increased by 50% compared to a standard dose on recovery time from deep neuromuscular block in elderly patients undergoing robot-assisted laparoscopic radical prostatectomy (RALP). Secondary objectives are to evaluate the different extubation time, time to exit from the operating room (OR), lenght of stay in post-anaesthesia care unit (PACU) and safety (hemodynamic parameters and respiratory function).

DETAILED DESCRIPTION:
An increasing percentage of elderly patients with localized prostate cancer undergo RALP, due to the higher safety and feasibility of this minimally invasive surgical option compared to standard open procedure. This procedure is performed under deep neuromuscular block (dNMB) in order to guarantee an adequate working space. Induction and maintenance of the dNMB require neuromuscular monitoring and adequate reversal at the end of the intervention to prevent postoperative residual curarization (PORC). Sugammadex is the most attractive strategy to titrate reversal according to NMB monitoring data and to ensure a complete recovery of muscle function before extubation. In elderly patients, the risk of PORC and related postoperative complications is higher. For these reasons, we hypothesize that a dose of sugammadex increased by 50% compared to a standard dose could significantly shorten neuromuscular recovery time, extubation time, OR discharge time and PACU length of stay in elderly patients undergoing RALP.

ELIGIBILITY:
Inclusion Criteria:

* patient's age ≥65years
* prostate cancer
* robot-assisted laparoscopic radical prostatectomy (RALP)

Exclusion Criteria:

* inability to obtain written informed consent
* history of significant liver, renal or pulmonary diseases
* current smoking
* chronic or acute alcoholism
* known or suspected neuromuscular disorders
* family history of malignant hyperthermia
* any pre-existing coagulopathy
* abnormal blood coagulation tests (including prothrombin time <70%; activated partial thromboplastin time >38 seconds and INR >1.20) or preoperative anticoagulant therapies
* BMI ≥30 Kg/m2
* known allergy or hypersensitivity to the drugs used in the study
* planned postoperative admission to intensive care unit.
* moderate neuromuscular block (TOF 1-3) at the end of surgery

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Neuromuscular recovery time | 5 minutes
  Time from the end of sugammadex administration to train-of-four (TOF)=1

SECONDARY OUTCOMES:
Time to extubation | 10 minutes
  Time from neuromuscular reversal (TOF=1) to extubation
Time to OR exit | 30 minutes
  Time from neuromuscular reversal (TOF=1) to exit from the operating room
PACU length of stay | 2 hours
  Duration of stay in the post-anaesthesia care unit
Hemodynamic parameters | up to discharge from post-anaesthesia care unit, an average of 2 hours
  Non-invasive blood pressure (mmHg) and heart rate (beats per minute) after sugammadex administration
Respiratory function | up to discarge from post-anaesthesia care unit, an average of 2 hours
  Peripheral oxygen saturation (percentage) and respiratory rate (breaths per minute) after sugammadex administration

CONTACTS AND LOCATIONS:
Overall Officials: Paola Aceto, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy